CLINICAL TRIAL: NCT00768378
Title: A Controlled Clinical Study to Evaluate the Safety and Efficacy of the BrainPort® Balance Device When Used to Improve Balance in Subjects With Peripheral Vestibular Dysfunction
Brief Title: Safety and Efficacy Study of BrainPort® Balance Device in Peripheral Vestibular Dysfunction.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wicab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WCB1-005; NIH: 2R44 DC004738
Record Dates: First submitted 2008-10-06; First posted 2008-10-08 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Vestibular Diseases; Gait Disorders
Keywords: Physical Therapy (Specialty); Balance dysfunction or disorder; Vestibular; Rehabilitation
MeSH Terms: conditions — Vestibular Diseases; Mobility Limitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perceived stimulation (Experimental): When subjects assigned to the perceived stimulation group increase the intensity of the stimulus, they will feel a tingling sensation on the tongue. The tingling will move on the tongue in relation to where the head/body moves.
  Interventions: Device: Training with the BrainPort balance device
- Subliminal stimulation (Experimental): When subjects assigned to the subliminal stimulation group increase the intensity of the stimulus, the device provides a stimulus that is below their conscious awareness, so they will not be able to perceive it. The stimulus will move on the tongue in relation to where the head/body moves.
  Interventions: Device: Training with the BrainPort balance device

INTERVENTIONS:
Device: Training with the BrainPort balance device — Subjects are randomly assigned to one of two groups, the perceived stimulation group or the subliminal stimulation group. Some of these devices provide a stimulus that you can feel. Others provide a stimulus that is below conscious awareness. We are conducting this study to determine if one type of stimulation is more effective than the other.
  Other Names: BrainPort Balance Device

SUMMARY:
The purpose of this study is to assess the safety and efficacy of the BrainPort balance device in improving balance and gait as measured by clinically accepted standardized balance assessments in subjects with peripheral vestibular dysfunction.

DETAILED DESCRIPTION:
Peripheral vestibular dysfunction can be caused by inner ear disorders, drug toxicity, neuritis, or a number of other causes. In the absence of a fully functional vestibular system, the brain often requires retraining to correctly utilize visual and proprioceptive cues to maintain postural stability. People with vestibular dysfunction experience multiple problems with posture control and movement, including an unsteady gait and various balance-related difficulties. These effects make it very difficult to walk in the dark or on uneven surfaces without risk of falling. They are typically referred for conventional vestibular therapy. Many patients improve with therapeutic intervention. Some patients reach a plateau and do not return to their previous level of function. The BrainPort balance device transmits head position information via electrotactile stimulation of the tongue. With training, patients learn to use the positional information to correct their balance.

Participants meeting the study criteria will be randomized to the perceived stimulation or subliminal stimulation group. All participants will be given baseline assessments of postural stability, balance, and subjective well being according to standardized tests. After completing the baseline assessments, each participant will be trained in the clinic using a standard training protocol with the BrainPort balance device. Each participant will participate in 6 clinical training sessions, over a period of 3 consecutive days. Upon completion of the clinic training sessions, participants will continue with a 7½ week period of home use. During this period, the participant will train with the device for 20 minutes 2 times per day and the clinicians will contact the participants weekly. At the end of the home training period (8 weeks from the beginning of the study), all participants will again undergo the tests given at baseline.

Following the data analysis, subjects that have completed the 8 week study and were originally assigned to the group with inferior results will be given the opportunity to use the device that showed superior results in the data analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of peripheral vestibular dysfunction by the following (within 12 months of study enrollment):

   1. Bilateral Vestibular Hypofunction (BVH)-Sinusoidal rotary chair results at least 2 SD below normal across the frequency range of 0.01 to 0.32 Hz, and at least 60 deg/s peak velocity.
   2. Unilateral Vestibular Hypofunction (UVH)-Bithermal caloric test results of > 25% unilateral weakness.
2. Minimum post 3 months diagnosis with residual balance problems.
3. Previously treated with conventional physical therapy, and discharged and/or reached a plateau.
4. Functional Ability:

   1. Able to ambulate independently or with an assistive device for 20 feet.
   2. Ability to stand independently for 2 minutes with no or minimal upper extremity support.
   3. Dynamic Gait Index ≤ 19/24.
5. Able to read and sign the informed consent form.
6. Fluent in English.
7. Willing and able to complete all testing, training, and follow-up evaluations required by the study protocol.

Exclusion Criteria:

1. Current oral health problems as determined by health questionnaire and an examination of the oral cavity.
2. Any medical condition that would interfere with performance on the assessments.
3. Known neuropathies of the tongue.
4. Prior exposure to BrainPort balance device.
5. History of seizures or epilepsy.
6. If female, pregnant. Subject must deny pregnancy and agree to use appropriate birth control to prevent pregnancy for the duration of the study.
7. People with implanted electrical medical devices (i.e. pacemaker, deep brain stimulator).
8. People currently taking any vestibular suppressant medication (i.e. barbiturates, benzodiazepines, betahistines or cortisone).
9. People with a previous diagnosis of a central nervous system lesion (e.g. stroke or brain injury).
10. Current diagnosis of any of the following:

    1. Bilateral areflexia (no response to ice water caloric testing bilaterally)
    2. Progressive neurological disease (such as Multiple Sclerosis)
    3. Cervicogenic dizziness
    4. Pre-syncope/syncope episodes
    5. Orthostatic hypotension
    6. Mood Disorders (such as Major Depression and Bipolar Disorder)
    7. Anxiety disorders
    8. Hydrops / Ménière's
11. Principal Investigator, in his or her medical judgment, does not believe the subject is a good candidate for the trial.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2008-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of the BrainPort balance device in improving balance and gait as measured by the Dynamic Gait Index (DGI) in subjects with documented peripheral vestibular dysfunction | Baseline and 8 weeks (end of study)

SECONDARY OUTCOMES:
To assess the safety of electrical stimulation of the tongue during the use of the BrainPort balance device in subjects with documented peripheral vestibular dysfunction. | Baseline and ongoing for the duration of the study (8 weeks).
To assess improvement in the Activities-specific Balance Confidence scale (ABC). | Baseline and 8 weeks (end of study)
To assess improvement in the Dizziness Handicap Inventory (DHI). | Baseline and 8 weeks (end of study)

CONTACTS AND LOCATIONS:
Overall Officials: James O. Phillips, PhD, Principal Investigator — University of Washington
Locations (17):
- United States (17):
  - England Physical Therapy, Los Angeles, California
  - South Valley Physical Therapy, PC, Centennial, Colorado
  - Sensory Therapeutics, Inc., Jupiter, Florida
  - NBC Rehabilitation, North Miami Beach, Florida
  - Atlanta Ear Clinic, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Elks Hearing & Balance Center, Boise, Idaho
  - Kansas University Medical Center, Kansas City, Kansas
  - Lahey Clinic, Burlington, Massachusetts
  - Missouri State University, Springfield, Missouri
  - New York Eye and Ear Infirmary, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Houston ENT Clinic, Houston, Texas
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Pacific Balance and Rehabilitation Clinic, Seattle, Washington
  - University of Washington School of Medicine, Seattle, Washington
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Background] Danilov YP, Tyler ME, Skinner KL, Hogle RA, Bach-y-Rita P. Efficacy of electrotactile vestibular substitution in patients with peripheral and central vestibular loss. J Vestib Res. 2007;17(2-3):119-30. PMID 18413905
- [Background] Bach-y-Rita P, W Kercel S. Sensory substitution and the human-machine interface. Trends Cogn Sci. 2003 Dec;7(12):541-6. doi: 10.1016/j.tics.2003.10.013. PMID 14643370
- [Background] Tyler M, Danilov Y, Bach-Y-Rita P. Closing an open-loop control system: vestibular substitution through the tongue. J Integr Neurosci. 2003 Dec;2(2):159-64. doi: 10.1142/s0219635203000263. PMID 15011268
- [Background] Bach-Y-Rita P. Emerging concepts of brain function. J Integr Neurosci. 2005 Jun;4(2):183-205. doi: 10.1142/s0219635205000768. PMID 15988797
- [Background] Danilov YP, Tyler ME, Skinner KL, Bach-y-Rita P. Efficacy of electrotactile vestibular substitution in patients with bilateral vestibular and central balance loss. Conf Proc IEEE Eng Med Biol Soc. 2006;Suppl:6605-9. doi: 10.1109/IEMBS.2006.260899. PMID 17959464
- [Background] Danilov Y, Tyler M. Brainport: an alternative input to the brain. J Integr Neurosci. 2005 Dec;4(4):537-50. doi: 10.1142/s0219635205000914. PMID 16385646